CLINICAL TRIAL: NCT06555042
Title: Investigation of VAP-1 Expression and Tissue Blood Flow by Combined [68Ga]DOTA-Siglec-9 and [15O]H2O PET-MRI in Patients With Small Bowel's Crohn's Disease
Brief Title: Investigation of VAP-1 Expression and Tissue Blood Flow by PET-MRI in Patients With Crohn's Disease
Acronym: VAP-PET
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Jukka Koffert, M.D., Ph.D., specialict in gastroenterology, Turku University Hospital
Other Study IDs: VARHA/4573/13.02.02/2024
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Crohn Disease; Inflammatory Bowel Diseases; Crohn Disease of Small Intestine; Crohn Colitis; Crohn's Ileocolitis; Crohn Disease in Remission
Keywords: Inflammatory Bowel Disease; Positron emission tomography; Crohn's disease; Vascular adhesion protein-1; Intestinal Perfusion
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples from endoscopy and whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, single center, imaging study. The CD patients with active disease will be assessed by [68Ga]Ga-DOTA-Siglec-9 and [15O]H2O PET/MRE. Patients with high clinical suspicion of small intestine's CD in outpatient gastroenterology clinic of Turku University Hospital will be recruited. The patients must fulfil the eligibility criteria and give their signed approvement prior to their enrolment into the study.

20 patients with high suspicion of active small bowels CD will be enrolled to being evaluated for potential participation in this study. In patients with diagnosed small bowels CD, PET-MRE will be repeated 3 months after the initial imaging (and based on clinical diagnostic started medication) to verify disease remission/inadequacy of the treatment.

Assessments for CD clinical disease activity will be performed at screening and [68Ga]Ga-DOTA-Siglec-9 and [15O]H2O PET/MRE assessments will be performed within a month for each patient.

After PET/MRE all patients can be treated according to patients' needs with immunosuppressive drugs. Follow-up visits are organized at after PET/MRE imaging at gastroenterology outpatient clinic.

DETAILED DESCRIPTION:
Patients with a strong suspicion of small bowel's CD after the colonoscopy and laboratory studies will be recruited to study protocol in the outpatient gastroenterology clinic of Turku University Hospital. After the signed informed consent patients will undergo combined [68Ga]Ga-DOTA-Siglec-9 and [15O]H2O PET/MRE, the MRE being part of their clinical diagnostics. If the MRE shows no signs/or mild inflammation of small intestine CD patients will be directed to small bowel capsule endoscopy (SBCE), which is routine in this clinical suspicion.

The patients will also have routine blood samples taken. A complete blood count (CBC), C-reactive protein (CRP), creatinine, alanine aminotransferase (ALAT), alkaline phosphatase (AFOS) and albumin will be analysed from each patient's blood sample, calprotectin and faecal microbiota will be analysed from stool. The tissue samples for (immuno)histological evaluation, proteome-wide mass spectrometry allowing sensitive site-specific detection of ADP-ribosylation and structural protein analysis will also be obtained in primary ileocolonoscopy (biopsies from the bowel wall).

Before the PET study starts, the patients will undergo screening procedures with physical examination, chemistry panel (electrolytes, creatinine, liver function), and acute phase reactants (ESR, CRP) and urine tests. In addition, serum/plasma biomarker sample, serum sample for soluble VAP-1 analysis, whole blood RNA sample, and whole blood DNA sample for gene variant analyses will be collected.

In the combined PET/MRE scanning the study subjects lay in the prone position on the PET scanner bed, and the area of interest (AOI) is positioned in the gantry and in the field of view.

[68Ga]Ga-DOTA-Siglec-9 and [15O]H2O PET/MRE imaging will be performed in the fasting state (at least 6 hours). The patients will be instructed to avoid caffeinated drinks during the last 24-hours before the study. A catheter will be inserted in an antecubital vein for injection of PET radiopharmaceutical. Another catheter will be inserted in the opposite radial or antecubital vein for blood sampling and the subjects will be placed in supine position in the PET/MRE scanner, arms next to the body. Ideally, urinary bladder should be empty before PET/MRE scan. The uptake of tracer will be measured using PET and MRE will be performed for anatomical reference.

After PET scans, the patients with CD will be treated and followed by gastroenterologist according to the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults between age 18-70
* Strong clinical suspicion of small bowel Crohn's disease
* Able and willing to give written informed consent and to comply with the study protocol

Exclusion Criteria:

* Pregnant or breast-feeding women
* Previous capsule retention
* X-ray investigations during preceding year
* Patients with metallic implants such as an electronic pacemaker or an implanted infusion pump
* Known stenosis of the GI-tract
* Evidence of significant uncontrolled concomitant diseases such as neurological, renal, hepatic, endocrine, or gastrointestinal disorders which, in the opinion of the Investigator, would preclude patient participation
* Is unable or unwilling to comply with the study protocol for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a strong suspicion of small bowel's CD after the colonoscopy and laboratory studies will be recruited to study protocol in the outpatient gastroenterology clinic of Turku University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
VAP-1 expression in the small bowel of patients with Crohn's disease | 18 months
  VAP-1 is expressed in the small bowel of patients with Crohn's disease and can be assessed by [68Ga]Ga-DOTA-Siglec-9 PET/MRE.

SECONDARY OUTCOMES:
VAP-1 immunohistochemistry | 18 months
  VAP-1 is expressed in the small bowel of patients with Crohn's disease and can be assessed by immunohistochemical staining of tissue biopsies.
Tissue perfusion | 18 months
  Intestinal blood flow is increased in inflamed small bowel and decreased in the late fibrosing stages of Crohn's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jukka Koffert, M.D., Ph.D, Principal Investigator — Turku University Hospital
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland